CLINICAL TRIAL: NCT03728790
Title: A Remote Postpartum (PP) Blood Pressure Surveillance and Reminder System for Hypertensive Disorders of Pregnancy: A Randomized Clinical Trial
Brief Title: Remote BP Monitoring in the PP Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Philips Healthcare (Industry); New York Presbyterian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAS0065
Record Dates: First submitted 2018-10-28; First posted 2018-11-02 (Actual); Results first posted 2020-09-28 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Hypertensive Disorder of Pregnancy
Keywords: hypertensive disorders of pregnancy; preeclampsia; gestational hypertension; HELLP
MeSH Terms: conditions — Toxemia; Pre-Eclampsia; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial with 2 arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Usual Care (No Intervention): Usual care group patients will be assigned to the usual care given to patients with hypertensive disorders of pregnancy at Columbia University Irving Medical Center (CUIMC). This involves a prescription for a blood pressure cuff if they do not already have one, with which they will be asked to measure their blood pressure twice per day. They will be asked to keep a log of their blood pressure measurements and to bring that log to their next provider visit.
- Remote Patient Monitoring (Experimental): Remote Patient Monitoring patients will use a Bluetooth-enabled blood pressure cuff, which will transmit blood pressure measurements via Bluetooth from the monitor to a tablet, which is able to be accessed by nurses staffing a remote clinical care center. Patients will also be prompted to answer surveys assessing symptoms of preeclampsia. The nurses will review measurements and survey results, which will be flagged in order of urgency. The measurements uploaded into the remote monitoring system will also be reviewed at the patient's next provider visit.
  Interventions: Device: Remote Patient Monitoring

INTERVENTIONS:
Device: Remote Patient Monitoring — Bluetooth-enabled blood pressure cuff to assess whether this technology helps providers collect more data regarding their patients' blood pressures in the postpartum period.
  Arms: Remote Patient Monitoring

SUMMARY:
The purpose of this study is to trial remote patient monitoring (RPM) in the postpartum hypertensive population in a randomized control design, with an aim to increase the number of blood pressure measurements taken during the fragile and under-monitored postpartum period and to thereby improve postpartum blood pressure control and reduce severe morbidity and mortality. The investigators plan to compare the number of blood pressures recorded in the first 10 days postpartum between patients who have been enrolled in an RPM trial to those who are being treated with the usual care.

DETAILED DESCRIPTION:
Many women develop high blood pressure as a complication of pregnancy. This high blood pressure can often take many weeks to resolve, and for some women it never resolves completely. If untreated, high blood pressure of pregnancy can lead to serious consequences, such as seizure or stroke. Unfortunately, because most women are sent home from the hospital just 2-3 days after having a baby, the best way of monitoring blood pressure at home is still unknown. Most women are given a prescription for a blood pressure cuff to use at home and an appointment to see their doctor at about one week after delivery to review their blood pressures, but many women have trouble checking their blood pressures, sometimes because they have a new baby at home and sometimes for other reasons like transportation or difficult social situations. Using a Bluetooth blood pressure monitoring system might help women have better blood pressure monitoring after they are discharged from the hospital after delivery, and therefore help to prevent some of the complications that can happen because of high blood pressure related to pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women
* Previous diagnosis of chronic hypertension, or antepartum diagnosis of hypertensive disorder of pregnancy (defined as documented blood pressure of ≥140 systolic or ≥90 diastolic on at least 2 occasions at least 4 hours apart)
* At least 18 years of age
* English or Spanish speakers

Exclusion Criteria:

* Non-English or Spanish speakers
* Women who are not planning on obtaining their postpartum follow up at CUIMC
* Women who are physically unable to hold or use the tablet
* Women who do not have a working phone
* Provider unwilling or unable to set up escalation pathway
* Women who reside outside of New York State
* Hypertension diagnosed postpartum

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2019-07-28 (Actual); Study Completion 2020-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Moroz, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Background] Goel A, Maski MR, Bajracharya S, Wenger JB, Zhang D, Salahuddin S, Shahul SS, Thadhani R, Seely EW, Karumanchi SA, Rana S. Epidemiology and Mechanisms of De Novo and Persistent Hypertension in the Postpartum Period. Circulation. 2015 Nov 3;132(18):1726-33. doi: 10.1161/CIRCULATIONAHA.115.015721. Epub 2015 Sep 28. PMID 26416810
- [Background] Creanga AA, Berg CJ, Syverson C, Seed K, Bruce FC, Callaghan WM. Pregnancy-related mortality in the United States, 2006-2010. Obstet Gynecol. 2015 Jan;125(1):5-12. doi: 10.1097/AOG.0000000000000564. PMID 25560097
- [Background] Levine LD, Nkonde-Price C, Limaye M, Srinivas SK. Factors associated with postpartum follow-up and persistent hypertension among women with severe preeclampsia. J Perinatol. 2016 Dec;36(12):1079-1082. doi: 10.1038/jp.2016.137. Epub 2016 Sep 1. PMID 27583396
- [Background] Bryant AS, Haas JS, McElrath TF, McCormick MC. Predictors of compliance with the postpartum visit among women living in healthy start project areas. Matern Child Health J. 2006 Nov;10(6):511-6. doi: 10.1007/s10995-006-0128-5. PMID 16807794
- [Background] Albini F, Xiaoqiu Liu, Torlasco C, Soranna D, Faini A, Ciminaghi R, Celsi A, Benedetti M, Zambon A, di Rienzo M, Parati G. An ICT and mobile health integrated approach to optimize patients' education on hypertension and its management by physicians: The Patients Optimal Strategy of Treatment(POST) pilot study. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:517-520. doi: 10.1109/EMBC.2016.7590753. PMID 28324932
- [Background] Sibai BM. Etiology and management of postpartum hypertension-preeclampsia. Am J Obstet Gynecol. 2012 Jun;206(6):470-5. doi: 10.1016/j.ajog.2011.09.002. Epub 2011 Sep 16. PMID 21963308
- [Background] Walters BN, Thompson ME, Lee A, de Swiet M. Blood pressure in the puerperium. Clin Sci (Lond). 1986 Nov;71(5):589-94. doi: 10.1042/cs0710589. PMID 3769407
- [Background] Clark SL, Belfort MA, Dildy GA, Englebright J, Meints L, Meyers JA, Frye DK, Perlin JA. Emergency department use during the postpartum period: implications for current management of the puerperium. Am J Obstet Gynecol. 2010 Jul;203(1):38.e1-6. doi: 10.1016/j.ajog.2010.02.033. Epub 2010 Apr 24. PMID 20417492
- [Background] Clapp MA, Little SE, Zheng J, Robinson JN. A multi-state analysis of postpartum readmissions in the United States. Am J Obstet Gynecol. 2016 Jul;215(1):113.e1-113.e10. doi: 10.1016/j.ajog.2016.01.174. PMID 27829570
- [Background] Al-Safi Z, Imudia AN, Filetti LC, Hobson DT, Bahado-Singh RO, Awonuga AO. Delayed postpartum preeclampsia and eclampsia: demographics, clinical course, and complications. Obstet Gynecol. 2011 Nov;118(5):1102-1107. doi: 10.1097/AOG.0b013e318231934c. PMID 21979459
- [Background] Bushnell C, McCullough LD, Awad IA, Chireau MV, Fedder WN, Furie KL, Howard VJ, Lichtman JH, Lisabeth LD, Pina IL, Reeves MJ, Rexrode KM, Saposnik G, Singh V, Towfighi A, Vaccarino V, Walters MR; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council for High Blood Pressure Research. Guidelines for the prevention of stroke in women: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 May;45(5):1545-88. doi: 10.1161/01.str.0000442009.06663.48. Epub 2014 Feb 6. PMID 24503673
- [Background] Wenger NK, Arnold A, Bairey Merz CN, Cooper-DeHoff RM, Ferdinand KC, Fleg JL, Gulati M, Isiadinso I, Itchhaporia D, Light-McGroary K, Lindley KJ, Mieres JH, Rosser ML, Saade GR, Walsh MN, Pepine CJ. Hypertension Across a Woman's Life Cycle. J Am Coll Cardiol. 2018 Apr 24;71(16):1797-1813. doi: 10.1016/j.jacc.2018.02.033. PMID 29673470
- [Background] Hirshberg A, Downes K, Srinivas S. Comparing standard office-based follow-up with text-based remote monitoring in the management of postpartum hypertension: a randomised clinical trial. BMJ Qual Saf. 2018 Nov;27(11):871-877. doi: 10.1136/bmjqs-2018-007837. Epub 2018 Apr 27. PMID 29703800
- [Background] Tully KP, Stuebe AM, Verbiest SB. The fourth trimester: a critical transition period with unmet maternal health needs. Am J Obstet Gynecol. 2017 Jul;217(1):37-41. doi: 10.1016/j.ajog.2017.03.032. Epub 2017 Apr 5. PMID 28390671
- [Background] ACOG Committee Opinion No. 736: Optimizing Postpartum Care. Obstet Gynecol. 2018 May;131(5):e140-e150. doi: 10.1097/AOG.0000000000002633. PMID 29683911
- [Background] Too G, Wen T, Boehme AK, Miller EC, Leffert LR, Attenello FJ, Mack WJ, D'Alton ME, Friedman AM. Timing and Risk Factors of Postpartum Stroke. Obstet Gynecol. 2018 Jan;131(1):70-78. doi: 10.1097/AOG.0000000000002372. PMID 29215510
- [Background] Gandapur Y, Kianoush S, Kelli HM, Misra S, Urrea B, Blaha MJ, Graham G, Marvel FA, Martin SS. The role of mHealth for improving medication adherence in patients with cardiovascular disease: a systematic review. Eur Heart J Qual Care Clin Outcomes. 2016 Oct 1;2(4):237-244. doi: 10.1093/ehjqcco/qcw018. PMID 29474713
- [Background] Arnhold M, Quade M, Kirch W. Mobile applications for diabetics: a systematic review and expert-based usability evaluation considering the special requirements of diabetes patients age 50 years or older. J Med Internet Res. 2014 Apr 9;16(4):e104. doi: 10.2196/jmir.2968. PMID 24718852
- [Background] Rhoads SJ, Serrano CI, Lynch CE, Ounpraseuth ST, Gauss CH, Payakachat N, Lowery CL, Eswaran H. Exploring Implementation of m-Health Monitoring in Postpartum Women with Hypertension. Telemed J E Health. 2017 Oct;23(10):833-841. doi: 10.1089/tmj.2016.0272. Epub 2017 May 5. PMID 28475431

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the inpatient postpartum service after delivery. Recruitment began on November 9, 2018. The last participant was recruited on July 10, 2019.
Period: Overall Study
Arm/Group | Usual Care | Remote Patient Monitoring
Started | 112 | 101
Completed | 112 | 101
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Remote Patient Monitoring | Total
Number analyzed (Participants) | 112 | 101 | 213
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [29 to 36] | 33 [28 to 36] | 33 [26 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 101 | 213
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 67 | 53 | 120
  Not Hispanic or Latino | 45 | 48 | 93
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 5 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 32 | 32 | 64
  White | 48 | 55 | 103
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 19 | 9 | 28
Multiparous [Count of Participants; unit: Participants] | 81 | 83 | 164
Married/Partnered [Number; unit: participants] | 76 | 89 | 165
Highest level of education [Count of Participants; unit: Participants] — Highest level of maternal education completed
  Participants
    Graduate School | 35 | 26 | 61
    College | 25 | 26 | 51
    Some college | 16 | 18 | 34
    High school | 26 | 27 | 53
    Some high school | 6 | 3 | 9
    Elementary school | 1 | 1 | 2
    Declined to answer | 3 | 0 | 3
Employment status [Count of Participants; unit: Participants]
  Employed | 75 | 66 | 141
  Unemployed | 33 | 30 | 63
  Self-employed | 4 | 5 | 9
Type of insurance [Count of Participants; unit: Participants]
  Public Insurance | 47 | 41 | 88
  Private Insurance | 65 | 60 | 125
Born outside of United States [Count of Participants; unit: Participants] | 54 | 49 | 103
Religion [Count of Participants; unit: Participants]
  Christian | 57 | 55 | 112
  Jewish | 4 | 7 | 11
  Muslim | 4 | 2 | 6
  Jehovah's Witness | 3 | 0 | 3
  Hindu | 0 | 2 | 2
  None | 37 | 34 | 71
  Other | 7 | 1 | 8
Type of prenatal care [Count of Participants; unit: Participants]
  Generalist | 62 | 55 | 117
  Maternal fetal medicine (MFM) | 45 | 43 | 88
  No prenatal care | 5 | 3 | 8
Smoking status [Count of Participants; unit: Participants]
  Current Smokers | 0 | 1 | 1
  Former Smokers | 6 | 5 | 11
Drug use status [Count of Participants; unit: Participants]
  Current users | 0 | 1 | 1
  Former users | 6 | 1 | 7
Time of initiation of prenatal care [Count of Participants; unit: Participants]
  First trimester | 84 | 82 | 166
  Second trimester | 24 | 15 | 39
  Third trimester | 1 | 2 | 3
  Unknown | 3 | 1 | 4
  No prenatal care | 0 | 1 | 1
Diabetes diagnosis [Count of Participants; unit: Participants]
  Type 1 Diabetes | 1 | 0 | 1
  Type 2 Diabetes | 4 | 1 | 5
  Gestational diabetes, diet controlled | 5 | 8 | 13
  Gestational diabetes, oral agents | 1 | 4 | 5
  Gestational diabetes, insulin | 7 | 3 | 10
Gestational age at delivery [Count of Participants; unit: Participants]
  20-23 6/7 weeks | 0 | 1 | 1
  24-27 6/7 weeks | 3 | 1 | 4
  28-33 6/7 weeks | 12 | 8 | 20
  34-36 6/7 weeks | 16 | 20 | 36
  37-38 6/7 weeks | 52 | 42 | 94
  39-40 6/7 weeks | 26 | 29 | 55
  >41 weeks | 3 | 0 | 3
Type of delivery [Count of Participants; unit: Participants]
  Cesarean Delivery | 56 | 57 | 113
  Spontaneous Vaginal Delivery | 53 | 43 | 96
  Forceps-assisted Vaginal Delivery | 3 | 1 | 4
Neonatal disposition [Count of Participants; unit: Participants]
  Fetal Demise | 1 | 0 | 1
  Neonatal Demise | 1 | 0 | 1
  Neonatal intensive care unit (NICU) admission | 28 | 19 | 47
Type of hypertension [Count of Participants; unit: Participants]
  Chronic Hypertension | 14 | 15 | 29
  Superimposed preeclampsia | 12 | 9 | 21
  Gestational Hypertension | 38 | 33 | 71
  Preeclampsia without severe features | 12 | 17 | 29
  Preeclampsia with severe features/HELLP Syndrome | 36 | 26 | 62
  Eclampsia | 0 | 1 | 1
Exposure to magnesium sulfate [Count of Participants; unit: Participants] | 44 | 34 | 78
Urgent antihypertensive medication antepartum or intrapartum [Count of Participants; unit: Participants] | 21 | 15 | 36
Discharged on antihypertensive medication [Count of Participants; unit: Participants] | 47 | 41 | 88

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure (BP) Surveillance Adherence
Description: Percentage of recommended twice-daily blood pressures reported between hospital discharge and first outpatient blood pressure assessment
Time Frame: Up to 14 days from delivery hospitalization discharge
Measure: Median (Full Range); unit: percentage of recommended BPs reported
Arm/Group | Usual Care | Remote Patient Monitoring
Number analyzed (Participants) | 112 | 101
percentage of recommended BPs reported | 0.0 [0.0 to 100.0] | 61.1 [0.0 to 92.3]

2. Secondary Outcome: Total Percentage of Elevated Blood Pressure Readings
Description: Of all blood pressure (BP) recordings collected per arm, the total percentage of those that were elevated will be reported. Elevated blood pressure defined as >/=140 systolic or >/=90 diastolic) by time of first outpatient blood pressure assessment (or 14 days from discharge, whichever came first).
Time Frame: Up to 14 days from delivery hospitalization discharge
Population: The analyzed population only includes participants who recorded at least one blood pressure at home after hospital discharge.
Measure: Number; unit: percentage of elevated BP readings
Arm/Group | Usual Care | Remote Patient Monitoring
Number analyzed (Participants) | 31 | 89
percentage of elevated BP readings | 37.52 | 49.6

3. Secondary Outcome: Number of Participants With Outpatient BP Assessment Within 14 Days
Description: Number of participants who had a documented outpatient BP assessment within 14 days of hospital discharge (excluding measurements taken at home)
Time Frame: Up to 14 days from delivery hospitalization discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Remote Patient Monitoring
Number analyzed (Participants) | 112 | 101
Participants | 69 | 59

4. Secondary Outcome: Percentage of Participants With Elevated BP After Discharge
Description: Incidence of elevated blood pressure (>140 systolic or >90 diastolic) at outpatient blood pressure assessment
Time Frame: Up to 14 days from delivery hospitalization discharge
Population: 1 participant in the Usual Care group attended but did not have BP recorded at outpatient visit. 2 participants in the Remote Patient Monitoring group attended but did not have BP recorded at outpatient visit.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | Remote Patient Monitoring
Number analyzed (Participants) | 68 | 57
percentage of participants | 27.9 | 24.5

5. Secondary Outcome: Number of Participants With Outpatient PP Assessment
Description: Number of participants who had an outpatient postpartum (PP) assessment
Time Frame: Up to 8 weeks from delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Remote Patient Monitoring
Number analyzed (Participants) | 112 | 101
Participants | 88 | 82

6. Secondary Outcome: Percentage of Participants With Elevated Blood Pressure at the Postpartum Visit
Description: Incidence of elevated blood pressure (>140 systolic or >90 diastolic) at the postpartum visit
Time Frame: Up to 8 weeks from delivery
Population: The analyzed population only includes participants who had an outpatient postpartum assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | Remote Patient Monitoring
Number analyzed (Participants) | 88 | 82
percentage of participants | 13.6 | 17.1

7. Secondary Outcome: Time to Medication Initiation
Description: Time to initiation of antihypertensive medications (in patients who were not on medications at time of discharge)
Time Frame: Up to 8 weeks from delivery
Population: The analyzed population only includes participants in each arm who were not on medications at the time of discharge.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Usual Care | Remote Patient Monitoring
Number analyzed (Participants) | 65 | 60
days | 6.5 [2.75 to 18] | 6.0 [3 to 13]

8. Secondary Outcome: Number of Participants Initiated on Antihypertensive Therapy After Hospital Discharge
Description: Number of participants discharged from delivery hospitalization without antihypertensive therapy, who were subsequently started on antihypertensive therapy
Time Frame: Up to 8 weeks from delivery
Population: The analyzed population only includes participants who were not on medications at the time of discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Remote Patient Monitoring
Number analyzed (Participants) | 65 | 60
Participants | 10 | 24

9. Secondary Outcome: Number of Participants Readmitted
Description: Number of participants who were readmitted after delivery hospitalization discharge
Time Frame: Up to 8 weeks from delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Remote Patient Monitoring
Number analyzed (Participants) | 112 | 101
Participants | 7 | 13

10. Secondary Outcome: Number of Participants With ED Visit
Description: Number of participants who had an Emergency Department (ED) visit after delivery hospitalization discharge
Time Frame: Up to 8 weeks from delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Remote Patient Monitoring
Number analyzed (Participants) | 112 | 101
Participants | 17 | 25

11. Secondary Outcome: Number of Participants Who Developed Preeclampsia-associated Complications
Description: Number of patients who experienced preeclampsia-related morbidity (eg: stroke, seizure, posterior reversible encephalopathy syndrome (PRES) , pulmonary edema, liver function abnormality, reversible cerebral vasoconstriction syndrome (RCVS) , renal insufficiency, thrombocytopenia) after delivery hospitalization discharge.
Time Frame: Up to 8 weeks from delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Remote Patient Monitoring
Number analyzed (Participants) | 112 | 101
Participants | 4 | 9

12. Secondary Outcome: Number of Participants Referred to Primary Care for Continued Blood Pressure Management
Description: Number of participants who require a referral to primary care physicians for continued blood pressure management after being discharged from obstetric care at the postpartum visit
Time Frame: Up to 8 weeks from delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Remote Patient Monitoring
Number analyzed (Participants) | 112 | 101
Participants | 31 | 38

13. Secondary Outcome: Score on the Modified Telemedicine Satisfaction and Usefulness Questionnaire (TSUQ)
Description: The modified TSUQ is an 18-item survey that will be used to measure patient satisfaction with remote blood pressure monitoring. Individuals score each of the items based on their satisfaction, with 1=strongly disagree to 5=strongly agree. The responses would then be used to calculate a mean score on the 5-point scale, with 5 indicating the most satisfaction.
Time Frame: Up to 8 weeks from delivery
Population: This questionnaire was not given to the Usual Care group since they did not participate in a telemedicine program.
  There were 52 respondents to the survey in the remote patient monitoring group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Remote Patient Monitoring
Number analyzed (Participants) | 0 | 52
score on a scale |  | 4.03 (0.95)

14. Secondary Outcome: Score on the Philips Program Start Survey and the Philips Program End Survey
Description: The Philips program start survey is a 4-question survey to gauge how patients relate to their care and their doctors prior to initiation of their blood pressure monitoring program. Individuals score each of the items based on the perception of their care, with 5 being best and 1 being worst. The responses would then be used to calculate a mean score on the 5-point scale, with 5 indicating the most satisfaction, and compared between the 2 groups. The Philips program end survey is a 6-question survey to gauge how patients related to their care and their doctors after the completion of their blood pressure monitoring program. Individuals score each of the items based on the perception of their care, with 5 being best and 1 being worst. The responses would then be used to calculate a mean score on the 5-point scale, with 5 indicating the most satisfaction, and compared between the 2 groups. The number reported is the average score for each group.
Time Frame: Baseline, program end (up to 8 weeks from delivery)
Population: The analyzed population only includes participants who completed both the Start Survey and the End Survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Remote Patient Monitoring
Number analyzed (Participants) | 61 | 42
score on a scale
  Baseline (Start Survey) | 4.77 (0.71) | 4.57 (2.23)
  Program End (End Survey) | 4.59 (0.82) | 4.55 (0.85)

15. Secondary Outcome: Communications
Description: Number of communications between patient and obstetric provider
Time Frame: Up to 14 days post delivery hospitalization discharge
Measure: Mean (Full Range); unit: Communications
Arm/Group | Usual Care | Remote Patient Monitoring
Number analyzed (Participants) | 112 | 101
Communications | 0.12 [0 to 2] | 0.57 [0 to 4]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through the end of the study period, which ended at the time of participants' postpartum visit or 8 weeks postpartum, whichever came first.
Arm/Group | Usual Care | Remote Patient Monitoring
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/101
Serious Adverse Events (participants affected / at risk) | 7/112 | 13/101
Other Adverse Events (participants affected / at risk) | 0/112 | 0/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=112) | Remote Patient Monitoring (N=101)
Readmission (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 13 (13) — This metric refers to hospital readmissions after delivery hospitalization discharge. This was also a secondary outcome metric of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT03728790/Prot_SAP_001.pdf